CLINICAL TRIAL: NCT05428657
Title: EC (Emotion and Cognition) Brain Program for Children With Special Education Needs in Primary School
Brief Title: EC Brain Program for Children With Special Education Needs
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Chan Sui-yin Agnes, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020.501-T
Record Dates: First submitted 2022-06-17; First posted 2022-06-23 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Neurodevelopmental Disorders
MeSH Terms: conditions — Neurodevelopmental Disorders

STUDY DESIGN:
Intervention Model Description: One group will be experimental and one group will active control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eye-tracking Training Group (Experimental): EC Brain After-school Program- computerised eye-tracking training program
  Interventions: Other: EC Brain After-school Program
- Conventional Training Group (Active Comparator): Conventional intervention program for special educational needs
  Interventions: Other: conventional intervention

INTERVENTIONS:
Other: EC Brain After-school Program — * Computerized Eye-tracking Attention and Impulse Control Training
  * Computerized Temporal Processing Training
  * Education on Relaxation, Stress Management and Healthy Balanced Diet
  Arms: Eye-tracking Training Group
Other: conventional intervention — Conventional cognitive training on their language and learning capacities (e.g., learning adjectives, logical reasoning, composition, reading words and story) and attention ability
  Arms: Conventional Training Group

SUMMARY:
Children with special education needs (SEN) (e.g., autism, attention-deficit/hyperactivity disorder, dyslexia) who are studying in the mainstream primary schools are commonly found to have difficulties in learning school materials, and controlling their emotion and behaviors in class. Such schooling problems are likely related to their deficient attention, self-control ability and language abilities. As a result, they will easily be stressful, losing confidence, or even be the target of bullying or discrimination. This project aims to evaluate a neuroscience based after-school training program, namely EC Brain Program, to improve academic performance, cognition (attention, self-control and language ability), behaviors and psychological health of primary school students with SEN. The EC Brain Program is composed of computerized training programs that were developed to enhance abilities of attention, self-control and temporal processing (i.e., a fundamental cognitive ability in mastering reading and language skills), and education on basic neuroscience knowledge and ways to enhance brain functions and psychological wellness, e.g., relaxation, stress management and balanced healthy diet. A total of 100 - 250 students with SEN from 10 ordinary primary schools will be recruited in 3-year period. They will be randomly assigned into two groups. Both groups will undergo pre- and post-assessments evaluating their academic performance, cognitive functions, saccadic eye movements, physical and mental health conditions before and after the training. Students in the group A will have to participate in the EC Brain after-school program, whereas students in the group B will join conventional intervention. It is an eight-month weekly program, 90 minutes per session. It is hypothesized that students who have joined the EC Brain Program will show greater extent of improvement in academic performance, behavioral problems, cognitive functions (e.g., attention, learning, self-control, language), saccadic eye movements and psychological wellness than those in the other group. The findings of present study will shed some light on the effectiveness and applicability of the EC Brain Program as a potential after-school neuropsychological intervention for students with SEN.

DETAILED DESCRIPTION:
Children with neurodevelopmental disorders are repeatedly found to have impairment in attention and self-control ability, which are part of executive functions and are largely mediated by the network among frontal, parietal and anterior cingulate brain regions. A recent review (Craig et al., 2016) suggested that ASD and ADHD share impairment in attention, response inhibition, working memory, flexibility, monitoring, fluency, and concept formation. In the review of Tarver and Hallahan (1974), children with SpLD were found to exhibit more distractibility on tasks, more impulsive and more hyperactive in a structured situation than typically developed children. Deficits in attention and self-control are highly associated with poorer school performance and more problem behaviors at school (Biederman et al., 2004; Riggs, Blair, Greenberg, 2010; Steinmayr, Ziegler, Träuble, 2010).

Eye gaze processing and temporal processing are two fundamental building blocks for higher cortical functions such as attention, memory, inhibitory control, language. Empirical research suggests that abnormal neurodevelopment of visual tracking correlates with the delayed maturation of functions in the frontal brain region, such as attention, inhibition and social communication (Johnson, 2001). In addition, children with SEN demonstrating abnormal cognitive functions or behaviours are found to have abnormal control of eye movement. For instance, atypical eye gazing at early stage of development is found to be related to attention deficit, joint attention and social functioning in ASD (Johnson, 2001). Abnormal eye movement is also evident in children with ADHD and reading disorder (Rommelse, Van der Stigchel & Sergeant, 2008). Increasing empirical research have been conducted to study the effectiveness of eye-tracking training in children with SEN. Powell et al. (2016) have conducted a computerized attention training to a group of ASD children using an eye-tracking system. After a training of 120 minutes within an average of 12 weeks, there was an improvement in visual sustained attention in a group of ASD children. Based on the similar concept, our research team has developed a gaze-contingent sustained attention and self-control training using the eye-tracking system. Our recent pilot study (Lee, Yeung, Sze, & Chan, 2021) revealed that 240-minute eye-tracking training for children with and without ADHD demonstrated significantly improved inhibitory control and mental flexibility after training, whereas children in the control group did not show significant changes.

Temporal processing underpinning all sensory and motor processing refers to how the nervous system processes time in the range of tens to hundreds of milliseconds. Temporal processing is a prerequisite condition for linguistic abilities (Schulte-Körne, Deimel, Bartling & Remschmidt, 1998) and highly associated with attention, memory and behavioural inhibition (Harrington & Haaland, 1999; Toplak, Dockstader, Tannock, 2006). Brain regions including basal ganglia, cerebellum, right parietal and dorsolateral prefrontal cortex play an important role in temporal processing (Mauk & Buonomano, 2004). Temporal processing deficits in visual or auditory modalities are repeatedly found among individuals with ASD, ADHD and SpLD. Kwakye et al., (2011) found that children with ASD demonstrated impaired auditory temporal processing as reflected by their higher threshold in the auditory temporal order judgment task comparing to typically developed children. Breier et al. (2003) found that children with ADHD or ADHD comorbid with reading disability showed a more pervasive deficit in perception of auditory temporal cues in nonspeech stimuli. Tallal (2004) and Merzenich et al. (2008) proposed that temporal processing deficit is basic deficit underlying the phonological and language difficulties of children with SpLD.

Meanwhile, it has been found that early intervention to improve auditory and visual temporal processing can have a significant positive impact on a child's learning. A systematic review (Loo et al., 2010) on the effectiveness of computer-based auditory training on processing non-speech and simple speech sounds has reported that some forms of training can improve children's phonological awareness skills (a fundamental skill for reading and verbal communication), whereas others may be effective in improving children's reading skills. Temple et al. (2003) conducted an empirical study and they found that 20 children with dyslexia demonstrated significantly improved oral language and reading performance after auditory processing training for an average of 27.9 training days, 100 min per day, 5 days per week. After the training, children with dyslexia showed increased activity in the left-sided brain regions, in which they showed hypo-activity compared to typically developed children before training. Wang, Liu, Xu (2019) also reported distinct effects of visual and auditory temporal processing training on reading and reading-related abilities in Chinese children with dyslexia. Children receiving 12 sessions, 3 to 4 times per week, 30-40 minutes per session of (1) auditory temporal processing training or (2) visual temporal processing training exhibited significantly improved reading and rapid naming ability. Yet, the control group with no specific training did not show such changes.

In view of the encouraging findings of eye tracking training and temporal processing training, the EC Brain after-school training program proposed in present study has thus incorporated these two forms of training for students with SEN. In addition to these two trainings, participating students are also educated on scientific lifestyle medicine methods to enhance their learning capacity and resilience against stress. They will be encouraged to develop a healthy life habit by practicing relaxation and stress management techniques and adopting a healthy balanced diet. According to WHO guidelines (2010), children aged 5-17 years old should accumulate at least 60 minutes of moderate-to vigorous-intensity physical activity daily, in order to improve physical and mental health. A traditional Chinese mind-body exercise, namely Neigong, involves gentle and calm movement and emphasizes on training self-awareness and concentration with a relaxed mind (Chan et al., 2008, 2011, 2013, 2015). It can be classified as a moderate intensity cardiovascular exercise and a relaxation exercise that primary school children can easily master. Research shows that one-month practice of the mind-body exercise can enhance self-control ability and memory function, and altered the corresponding brain activity level of children with ASD (Chan et al., 2008, 2013, 2015). Clinical observation also showed better control of temper and impulsive acts, and higher resilience against stressors after regular practice of Neigong in children with SEN. A healthy balanced diet according to MyPlate is the nutrition guide published by the United States Department of Agriculture (USDA). MyPlate suggests intake of healthy food at a specified balanced proportion: Whole grains (30%), Vegetables and Fruits (50%), and Protein (20%). For the Protein category, more emphasis is put on a higher intake of plant-based protein (e.g., seeds, beans, nuts). Children with ASD adopting the balanced healthy diet showed significantly enhanced cognitive flexibility, impulse control and planning ability, reduced social communication problem and repetitive behaviors, and increased EEG brain activity (Chan, et al., 2012a).

The primary objective of the present study is to examine the effectiveness and applicability of a neuroscience-based after-school EC Brain Program in improving academic performance, cognition, saccadic eye movements, behaviors and psychological health of 100-250 Chinese students with SEN from 10 ordinary local primary schools. It is hypothesized that students joining EC Brain Program will demonstrate greater extent of improvement in academic performance, attention, self-control, language ability, and saccadic eye movements, greater reduction in behavioral problems and better psychological well-being after training. In contrast, children in the conventional training group will not have similar extent of improvements as the EC Brain group.

ELIGIBILITY:
Inclusion Criteria:

* primary school Chinese students with SEN (e.g., Autism Spectrum Disorders, Attention-Deficit/Hyperactivity Disorders, Specific Learning Disorders)
* aged between 6 to 12 years
* with formal diagnosis of neurodevelopmental disorders by psychiatrist or clinical / educational psychologist

Exclusion Criteria:

・students with mental disabilities, significant physical disability, or history of other neurological or psychiatric disorder or brain injury

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 328 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Wechsler Intelligence Scale for Children, 4th edition (Hong Kong) | 10 minutes
  It is an intellectual functioning test. The short-form comprising four subtests will adopted to estimate full scale IQ. The scaled scores of each subtest will be computed, ranging from 1 to 19, where higher scores indicate better performance.
Hong Kong List Learning Test | 10 minutes
  It is a memory test which composes of three learning trials of 16 Chinese words, and two delayed recall trials. The score ranges from 0 to 16 in each trial, where higher scores indicate better performance.
Conners' Continuous Performance Test | 15 minutes
  Attention Test
Shape Trail Test | 10 minutes
  Attention Test and flexibility
Tinkertoy Test | 5 minutes
  Frontal functioning test
Interview and Questionnaires for Parents and Teachers | 20 minutes
  structured interview to collect information about students' behaviors at home and in class
saccadic testing | 30 minutes
  Saccadic eye movements will be measured during the tests included but not limited to pro-saccade and anti-saccade tasks, the rapid digit and letter naming tasks, the Chinese and English passage reading, and the Corsi task

CONTACTS AND LOCATIONS:
Overall Officials: Agnes SY Chan, Professor, Principal Investigator — Chinese University of Hong Kong
Locations (3):
- The Chinese University of Hong Kong, Hong Kong, China
- Hong Kong (2):
  - Neuropsychology Laboratory, Department of Psychology, The Chinese University of Hong Kong, Hong Kong
  - The Chinese University of Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
The investigator do not plan to share Individual Participant Data. It is because this study is funded by a private funding source, the data are belonged to that source. So, sharing IPD is not available.

REFERENCES:
- [Result] Biederman J, Monuteaux MC, Doyle AE, Seidman LJ, Wilens TE, Ferrero F, Morgan CL, Faraone SV. Impact of executive function deficits and attention-deficit/hyperactivity disorder (ADHD) on academic outcomes in children. J Consult Clin Psychol. 2004 Oct;72(5):757-66. doi: 10.1037/0022-006X.72.5.757. PMID 15482034
- [Result] Breier JI, Fletcher JM, Foorman BR, Klaas P, Gray LC. Auditory temporal processing in children with specific reading disability with and without attention deficit/hyperactivity disorder. J Speech Lang Hear Res. 2003 Feb;46(1):31-42. doi: 10.1044/1092-4388(2003/003). PMID 12647886
- [Result] Chan AS, Cheung MC, Sze SL, Leung WW, Shi D. Shaolin dan tian breathing fosters relaxed and attentive mind: a randomized controlled neuro-electrophysiological study. Evid Based Complement Alternat Med. 2011;2011:180704. doi: 10.1155/2011/180704. Epub 2010 Sep 22. PMID 20976126
- [Result] Chan AS, Han YM, Sze SL, Lau EM. Neuroenhancement of Memory for Children with Autism by a Mind-Body Exercise. Front Psychol. 2015 Dec 11;6:1893. doi: 10.3389/fpsyg.2015.01893. eCollection 2015. PMID 26696946
- [Result] Chan AS, Sze SL, Han YM, Cheung MC. A chan dietary intervention enhances executive functions and anterior cingulate activity in autism spectrum disorders: a randomized controlled trial. Evid Based Complement Alternat Med. 2012;2012:262136. doi: 10.1155/2012/262136. Epub 2012 May 14. PMID 22666288
- [Result] Chan, A.S., Sze, S.L., & Shi, D. (2008). Traditional Chinese mind-body exercises improve self control ability of an adolescent with Asperger's disorder. Journal of Psychology in Chinese Societies, 9, 225-239.
- [Result] Chan AS, Sze SL, Siu NY, Lau EM, Cheung MC. A chinese mind-body exercise improves self-control of children with autism: a randomized controlled trial. PLoS One. 2013 Jul 10;8(7):e68184. doi: 10.1371/journal.pone.0068184. Print 2013. PMID 23874533
- [Result] Chan AS, Wong QY, Sze SL, Kwong PP, Han YM, Cheung MC. A Chinese Chan-based mind-body intervention for patients with depression. J Affect Disord. 2012 Dec 15;142(1-3):283-9. doi: 10.1016/j.jad.2012.05.018. Epub 2012 Jul 25. PMID 22840618
- [Result] Chan AS, Wong QY, Sze SL, Kwong PP, Han YM, Cheung MC. A Chinese chan-based mind-body intervention improves sleep on patients with depression: a randomized controlled trial. ScientificWorldJournal. 2012;2012:235206. doi: 10.1100/2012/235206. Epub 2012 Apr 30. PMID 22623888
- [Result] Craig F, Margari F, Legrottaglie AR, Palumbi R, de Giambattista C, Margari L. A review of executive function deficits in autism spectrum disorder and attention-deficit/hyperactivity disorder. Neuropsychiatr Dis Treat. 2016 May 12;12:1191-202. doi: 10.2147/NDT.S104620. eCollection 2016. PMID 27274255
- [Result] Harrington DL, Haaland KY. Neural underpinnings of temporal processing: a review of focal lesion, pharmacological, and functional imaging research. Rev Neurosci. 1999;10(2):91-116. doi: 10.1515/revneuro.1999.10.2.91. PMID 10658954
- [Result] Johnson MH. Functional brain development in humans. Nat Rev Neurosci. 2001 Jul;2(7):475-83. doi: 10.1038/35081509. No abstract available. PMID 11433372
- [Result] Kwakye LD, Foss-Feig JH, Cascio CJ, Stone WL, Wallace MT. Altered auditory and multisensory temporal processing in autism spectrum disorders. Front Integr Neurosci. 2011 Jan 5;4:129. doi: 10.3389/fnint.2010.00129. eCollection 2011. PMID 21258617
- [Result] Lee TL, Yeung MK, Sze SL, Chan AS. Computerized Eye-Tracking Training Improves the Saccadic Eye Movements of Children with Attention-Deficit/Hyperactivity Disorder. Brain Sci. 2020 Dec 21;10(12):1016. doi: 10.3390/brainsci10121016. PMID 33371236
- [Result] Lee TL, Yeung MK, Sze SL, Chan AS. Eye-Tracking Training Improves Inhibitory Control in Children with Attention-Deficit/Hyperactivity Disorder. Brain Sci. 2021 Mar 2;11(3):314. doi: 10.3390/brainsci11030314. PMID 33801559
- [Result] Loo JH, Bamiou DE, Campbell N, Luxon LM. Computer-based auditory training (CBAT): benefits for children with language- and reading-related learning difficulties. Dev Med Child Neurol. 2010 Aug;52(8):708-17. doi: 10.1111/j.1469-8749.2010.03654.x. Epub 2010 Mar 29. PMID 20370814
- [Result] Mauk MD, Buonomano DV. The neural basis of temporal processing. Annu Rev Neurosci. 2004;27:307-40. doi: 10.1146/annurev.neuro.27.070203.144247. PMID 15217335
- [Result] Merzenich M, Wright B, Jenkins W, Xerri C, Byl N, Miller S, Tallal P. Cortical plasticity underlying perceptual, motor, and cognitive skill development: implications for neurorehabilitation. Cold Spring Harb Symp Quant Biol. 1996;61:1-8. No abstract available. PMID 9246429
- [Result] Powell G, Wass SV, Erichsen JT, Leekam SR. First evidence of the feasibility of gaze-contingent attention training for school children with autism. Autism. 2016 Nov;20(8):927-937. doi: 10.1177/1362361315617880. Epub 2016 Feb 9. PMID 26862085
- [Result] Riggs NR, Blair CB, Greenberg MT. Concurrent and 2-year longitudinal relations between executive function and the behavior of 1st and 2nd grade children. Child Neuropsychol. 2003 Dec;9(4):267-76. doi: 10.1076/chin.9.4.267.23513. PMID 14972705
- [Result] Rommelse NN, Van der Stigchel S, Sergeant JA. A review on eye movement studies in childhood and adolescent psychiatry. Brain Cogn. 2008 Dec;68(3):391-414. doi: 10.1016/j.bandc.2008.08.025. Epub 2008 Oct 2. PMID 18835079
- [Result] Schulte-Korne G, Deimel W, Bartling J, Remschmidt H. Role of auditory temporal processing for reading and spelling disability. Percept Mot Skills. 1998 Jun;86(3 Pt 1):1043-7. doi: 10.2466/pms.1998.86.3.1043. PMID 9656305
- [Result] Steinmayr, R., Ziegler, M., & Träuble, B. (2010). Do intelligence and sustained attention interact in predicting academic achievement?. Learning and Individual Differences, 20(1), 14-18.
- [Result] Tarver S. G., & Hallahan, D. P. (1974). Attention deficits in children with learning disabilities: a review. Journal of Learning Disabilities, 7, 560-569.
- [Result] Tallal P. Improving language and literacy is a matter of time. Nat Rev Neurosci. 2004 Sep;5(9):721-8. doi: 10.1038/nrn1499. PMID 15322530
- [Result] Temple E, Deutsch GK, Poldrack RA, Miller SL, Tallal P, Merzenich MM, Gabrieli JD. Neural deficits in children with dyslexia ameliorated by behavioral remediation: evidence from functional MRI. Proc Natl Acad Sci U S A. 2003 Mar 4;100(5):2860-5. doi: 10.1073/pnas.0030098100. Epub 2003 Feb 25. PMID 12604786
- [Result] Toplak ME, Dockstader C, Tannock R. Temporal information processing in ADHD: findings to date and new methods. J Neurosci Methods. 2006 Feb 15;151(1):15-29. doi: 10.1016/j.jneumeth.2005.09.018. Epub 2005 Dec 27. PMID 16378641
- [Result] Tuso PJ, Ismail MH, Ha BP, Bartolotto C. Nutritional update for physicians: plant-based diets. Perm J. 2013 Spring;17(2):61-6. doi: 10.7812/TPP/12-085. PMID 23704846
- [Result] Wang LC, Liu D, Xu Z. Distinct effects of visual and auditory temporal processing training on reading and reading-related abilities in Chinese children with dyslexia. Ann Dyslexia. 2019 Jul;69(2):166-185. doi: 10.1007/s11881-019-00176-8. Epub 2019 Jan 22. PMID 30671864
- [Result] Zhao Q, Guo Q, Li F, Zhou Y, Wang B, Hong Z. The Shape Trail Test: application of a new variant of the Trail making test. PLoS One. 2013;8(2):e57333. doi: 10.1371/journal.pone.0057333. Epub 2013 Feb 20. PMID 23437370
- [Derived] Chan AS, Leung PY, Pang TW, Sze SL. Eye-tracking training improves visuospatial working memory of children with attention-deficit/hyperactivity disorder and autism spectrum disorder. Autism Res. 2024 Nov;17(11):2244-2260. doi: 10.1002/aur.3238. Epub 2024 Oct 4. PMID 39364754
- [Derived] Chan AS, Sze SL, Cheung MC. Temporal processing tele-intervention improves language, attention, and memory in children with neurodevelopmental disorders. Digit Health. 2023 Sep 28;9:20552076231203900. doi: 10.1177/20552076231203900. eCollection 2023 Jan-Dec. PMID 37780065